CLINICAL TRIAL: NCT06418425
Title: EPPIC Trial: Exercise Program and Protein Intake Counselling for Frailty Prevention in Singapore
Brief Title: Exercise Program and Protein Intake Counselling for Frailty Prevention in Singapore
Acronym: EPPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group Polyclinics (Other Government)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/00860; EPHF-C/2023/POV/S/4 (Other Grant/Funding Number: NHG ENHANCED POPULATION HEALTH FUND (EPHF))
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-05

CONDITIONS: Frailty
Keywords: frailty; pre-frailty; primary care; exercise; high protein diet; nutrition
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants meeting the eligibility criteria, will be approached by the care coordinator. If interested in participating, they will be referred to the research team member for recruitment and consent will be taken. Participants will then be randomly assigned to "intervention" or "usual care" parallel arms. Randomisation of participants will be done on 1:1 allocation to intervention or usual care using block randomisation. Allocation will be concealed using opaque envelopes.
Who Masked: Outcomes Assessor
Masking Description: Research coordinator who assesses the outcomes will be blinded. This clinical research coordinator is different from the one taking the informed consent and performing the randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants randomly assigned to the intervention group will be taught specific resistance, balance and aerobic exercises by the care co-ordinator and participants will receive a leaflet with pictorial guide on the home-based exercise regime. The participants will be given a monitoring log to record the date and frequency of exercise they do. The participants will be advised to consume adequate protein and they will also receive another leaflet on protein consumption as part of a balanced diet.
  Interventions: Behavioral: counselling on home-based exercise program and dietary protein intake
- Usual Care (No Intervention): Participants in the control group will receive usual care at the polyclinic which does not include counselling on dietary protein intake and home-based exercise program.

INTERVENTIONS:
Behavioral: counselling on home-based exercise program and dietary protein intake — Participants in the intervention group will be on a home-based exercise program and go through counselling on dietary protein intake with the aim of achieving prevention of frailty status. Participants will be required to attend the 3 study visits throughout the study period. Research procedures include physical measurements (eg. Weight, height, waist and hip circumference, calf circumference, hand grip strength, blood pressure, short physical performance battery tests), administration of questionnaires on sociodemographics, physical activity, dietary habits, smoking, alcohol, health conditions, health-related quality of life, clinical frailty status and sarcopenia screening. At three months and twelve months, the intervention group participants will see the care coordinators who will check their compliance to the exercise programme and high protein diet, reinforce the interventions.
  Arms: Intervention

SUMMARY:
This is a randomized controlled trial that is designed to study the effectiveness of home-based exercise program and high dietary protein counselling in preventing frailty among elderly in Singapore primary care setting.

DETAILED DESCRIPTION:
The investigators are studying the elderly population who have prefrailty (Fried Frailty). Participants include those who are: a) Aged 65 to 100 years old b) screened CFS 3-4. Patients will be approached via phone call by care coordinators, as part of the routine care. As part of the routine care to our chronic patients, care coordinators identify eligible patients for annual screening to update personal particulars/ cancer screening and vaccination statuses as per the Healthier SG program before patient's chronic disease appointment. Also as part of the routine care, care coordinators will screen for CFS 3 and 4 patients over the phone. Patients who fulfil CFS 3 and 4 will be arranged to have a physical consultation with care coordinators on their day of prescheduled visit in the clinic. Patients meeting the eligibility criteria for the study, will be approached by the care coordinator to ask for research interest. If interested in participating, patients will be referred to the research team member for recruitment and consent will be taken. Participants will then be randomly assigned to "intervention" or "usual care" parallel arms. Randomisation of participants will be done on 1:1 allocation to intervention or usual care by a simple randomisation procedure. Participants randomly assigned to the usual care group will receive normal primary care, including dietitian and physiotherapy services if needed. Intervention participants will receive the described intervention on top of usual care. Intervention participants will be taught specific resistance and balance exercises and participants will receive a leaflet with pictorial guide on the home based exercise regime. The participants will be advised to consume adequate protein and participants will also receive another leaflet on protein consumption as part of a balanced diet. At the 3 month and 12 month mark, participants in the intervention group will see the care coordinator who will assess compliance and re-enforce the exercise regime and dietary protein intake counselling, and check for any difficulties faced.

ELIGIBILITY:
Inclusion Criteria:

* 65 - 100 years old
* Community dwelling
* On chronic disease follow up with polyclinic
* Ability to communicate in English or Mandarin
* Able to understand the study and give consent

Exclusion Criteria:

* Individuals with existing dietitian/ physiotherapy intervention (Individuals who are already seeing dietitian for special delivery requirements, or seeing physiotherapist for musculoskeletal exercises for specific condition or injury)
* Institutionalized individuals
* Individuals with significant medical conditions limiting their physical activity or high protein diet, such as severe heart conditions, recent strokes, active malignancy, chronic kidney disease stage 3-5 etc.
* Terminal illness with life expectancy < 12 months
* severe audiovisual impairment
* Not able to communicate in English or Mandarin
* Pregnant women ( as population involves participants beyond childbearing age, investigators do not expect to include pregnant women in this study)

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-18 (Estimated)

PRIMARY OUTCOMES:
Repeated Chair Rise Test | Baseline, 3 months, 12 months
  Measured with repeated chair rise test which is a functional performance frailty metric. As the intervention is more exercise based, the primary outcome will be able to capture the changes brought about by the intervention.

SECONDARY OUTCOMES:
Clinical Frailty Scale (CFS) | Baseline, 3 months, 12 months
  The CFS is a scale that ranges from 1 to 9, with each number representing a different level of frailty, depending on the physical activity level, fatigue level and functional level of the participant. The care-coordinator will assign a CFS score after a brief assessment of the participant. Additionally, the participant will also completed a self-rated CFS questionnaire (CFS-self) that will rate their CFS level. CFS 1 is very fit, with progressive frailty status down the scale to maximum CFS 9 for terminally ill.
Short Physical Performance Battery (SPPB) | Baseline, 3 months, 12 months
  The SPPB (score range 0-12) consists of chair-stand, gait speed and standing balance. In the balance test, the participant will be made to stand in three different feet positions (side-by-side, semi-tandem, tandem) for 10 seconds each and will be scored for how long they are able to hold that position. The gait speed test will score the participants based on how long they take to walk three meters. Lastly, the chair rise test will score the participants on how long they take to complete five raises from a seated position in a chair.
Health-related Quality of life | Baseline, 3 months, 12 months
  Measured by the EuroQoL 5 Dimensions - 5L (EQ5D-5L) and the EuroQoL 5 Visual Analogue Scale (EQ5D-VAS). The EQ5D-5L consists of two components, the first component is the healthstate Utility Index (UI). It measures five dimensions of health-related quality of life (mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression) on a five-point severity scale (no problems, slight problems, moderate problems, severe problems and extreme problems). The Singapore time trade-off values will be used to convert the information into UI scores, with -0.790 being the worst health state and 1.000 being the best health state. The second component of the EQ5D is the visual analogue scale (VAS) which consists of a scale from 0 to 100. It assesses self-perceived global levels of health, with 0 representing the worst imaginable health state and 100 the best imaginable health state.
Sarcopenia | Baseline, 3 months, 12 months
  According to the Asian Work Group of Sarcopenia (AWGS) 2019 criteria, which is SARC-Calf more than or equal to 11 and poor handgrip strength (<28kg for men and <18kg for women). The SARC-Calf is a combination of assessments for the SARC-F questionnaire and calf-circumference. The SARC-F questionnaire has 5 items measuring self-reported strength, assistance in walking, difficulty rising from a chair, difficulty in climbing stairs, and falls in the past year. Each item requires a response of "None" or "Some" or "Great difficulty", except for the last item on falls which has responses of "None" or "1-3 falls" or "4 or more falls". The calf circumference measures the maximum value of both calves using a non-elastic tape, with a cut-off of <34cm for men and <33cm for women for sarcopenia case finding. Each item of the SARC-Calf is scored 0-2 and the items are summed together to give a total score.
Physical activity | Baseline, 3 months, 12 months
  Measured by International physical activity questionnaire (IPAQ). 3.3 METs for low level, 4.0 METs for moderate level, and 8.0 METs high level of physical activity.
Dietary Protein Intake | Baseline, 3 months, 12 months
  Measured by 24-hour dietary recall and food frequency on protein sources. Participants will be asked to recall the food or drink they consumed the previous day in detail. The information collected will be analyzed to quantify daily protein intake in grams. Additionally, participants will be asked to complete a brief food frequency questionnaire on various protein sources.

CONTACTS AND LOCATIONS:
Overall Officials: Liew Pui Mun Doctor, MBBS, Principal Investigator — National Healthcare Group Polyclinic
Locations (1):
- Ang Mo Kio Polyclinic, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra-Prat M, Sist X, Domenich R, Jurado L, Saiz A, Roces A, Palomera E, Tarradelles M, Papiol M. Effectiveness of an intervention to prevent frailty in pre-frail community-dwelling older people consulting in primary care: a randomised controlled trial. Age Ageing. 2017 May 1;46(3):401-407. doi: 10.1093/ageing/afw242. PMID 28064172
- [Background] Travers J, Romero-Ortuno R, Bailey J, Cooney MT. Delaying and reversing frailty: a systematic review of primary care interventions. Br J Gen Pract. 2019 Jan;69(678):e61-e69. doi: 10.3399/bjgp18X700241. Epub 2018 Dec 3. PMID 30510094